CLINICAL TRIAL: NCT04978519
Title: Evaluation of the Effectiveness of Cryotherapy for the Treatment of Prostate Cancer
Brief Title: Effectiveness of Cryotherapy Study for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Hang Yee, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2020.018
Record Dates: First submitted 2021-07-22; First posted 2021-07-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Focal therapy; Cryotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryotherapy (Experimental): Cryotherapy achieves a temperature averaging -40°C. Through the transperineal insertion of treatment probes, it exerts its effect through freezing of tissue and vascular injury, leading to destruction of cancer tissue.
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Cryotherapy — Cryotherapy is administered by using perineal needles, placed under ultrasound guidance to freeze the target tissue.

SUMMARY:
This is a single-centre prospective, non-randomized trial to investigate the efficacy of cryotherapy in patients with localized prostate cancer.The aim of study is to investigate the safety profile of cryotherapy in the treatment of prostate cancer and to evaluate the oncological control of prostate cancer by means of cryotherapy focal treatment.

DETAILED DESCRIPTION:
Conventional treatment options for localized prostate cancer include prostatectomy, radiotherapy and active surveillance. However, prostatectomy and radiotherapy carry certain degree of morbidity, including the risks of urinary incontinence, erectile dysfunction and injury to the structures in the proximity. Active surveillance carries the risk of disease progression and psychological distress to the patients. Focal therapy employs the concept of only destroying the significant lesion, resulting in disease cure and improved functional outcome. Among the different options of focal therapy, cryotherapy is one of the most commonly employed energy sources. It exerts its effect through freezing of tissue and vascular injury, leading to destruction of cancer tissue. Our study aims at assess the safety and effectiveness of such treatment in prostate cancer management

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 40 - 85 years
* Visible index lesion(s) on MRI
* Found to have localized prostate cancer after MRI-USG fusion targeted biopsy:

  1. Clinical tumour stage <= T2, or
  2. Gleason score <= 7, or
  3. PSA <= 20 ng/ml

Exclusion Criteria:

* Patients unfit for contrast MRI exam
* Patients with active urinary tract infection
* Patients with bladder pathology including bladder stone and bladder cancer
* Patients with urethral stricture
* Patients with neurogenic bladder and/or sphincter abnormalities
* Patients who fail to give informed consent

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only man will develop prostate cancer
Enrollment: 16 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Oncological outcome-mpMRI prostate | 6 months
  Oncological outcome after cryotherapy treatment, as defined by mpMRI prostate

SECONDARY OUTCOMES:
Oncological Outcomes after cryotherapy | 12 months
  Oncological outcome after cryotherapy treatment, as defined by mpMRI
Functional outcome after cryotherapy | 6 months and 12 months
  Change in scores in EPIC-26 questionnaires
Complication after study intervention | 30 days
  Post treatment complication
Oncological outcome-Biopsy | 12 months
  Presence of histologically proven prostate cancer recurrence on biopsy in suspicious cases
Prostate Specific Antigen change | 3 months, 6 months, 9 months, 12 months
  PSA change after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hang YEE, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stamey TA, Caldwell M, McNeal JE, Nolley R, Hemenez M, Downs J. The prostate specific antigen era in the United States is over for prostate cancer: what happened in the last 20 years? J Urol. 2004 Oct;172(4 Pt 1):1297-301. doi: 10.1097/01.ju.0000139993.51181.5d. PMID 15371827
- [Background] Klotz L, Vesprini D, Sethukavalan P, Jethava V, Zhang L, Jain S, Yamamoto T, Mamedov A, Loblaw A. Long-term follow-up of a large active surveillance cohort of patients with prostate cancer. J Clin Oncol. 2015 Jan 20;33(3):272-7. doi: 10.1200/JCO.2014.55.1192. Epub 2014 Dec 15. PMID 25512465
- [Background] Kaye DR, Qi J, Morgan TM, Linsell S, Ginsburg KB, Lane BR, Montie JE, Cher ML, Miller DC; Michigan Urological Surgery Improvement Collaborative. Pathological upgrading at radical prostatectomy for patients with Grade Group 1 prostate cancer: implications of confirmatory testing for patients considering active surveillance. BJU Int. 2019 May;123(5):846-853. doi: 10.1111/bju.14554. Epub 2018 Oct 15. PMID 30248225
- [Background] Lindner U, Trachtenberg J, Lawrentschuk N. Focal therapy in prostate cancer: modalities, findings and future considerations. Nat Rev Urol. 2010 Oct;7(10):562-71. doi: 10.1038/nrurol.2010.142. Epub 2010 Sep 14. PMID 20842187
- [Background] Donaldson IA, Alonzi R, Barratt D, Barret E, Berge V, Bott S, Bottomley D, Eggener S, Ehdaie B, Emberton M, Hindley R, Leslie T, Miners A, McCartan N, Moore CM, Pinto P, Polascik TJ, Simmons L, van der Meulen J, Villers A, Willis S, Ahmed HU. Focal therapy: patients, interventions, and outcomes--a report from a consensus meeting. Eur Urol. 2015 Apr;67(4):771-7. doi: 10.1016/j.eururo.2014.09.018. Epub 2014 Oct 1. PMID 25281389
- [Background] Babaian RJ, Donnelly B, Bahn D, Baust JG, Dineen M, Ellis D, Katz A, Pisters L, Rukstalis D, Shinohara K, Thrasher JB. Best practice statement on cryosurgery for the treatment of localized prostate cancer. J Urol. 2008 Nov;180(5):1993-2004. doi: 10.1016/j.juro.2008.07.108. Epub 2008 Sep 25. No abstract available. PMID 18817934
- [Background] Ward JF, Jones JS. Focal cryotherapy for localized prostate cancer: a report from the national Cryo On-Line Database (COLD) Registry. BJU Int. 2012 Jun;109(11):1648-54. doi: 10.1111/j.1464-410X.2011.10578.x. Epub 2011 Oct 28. PMID 22035200